CLINICAL TRIAL: NCT05406024
Title: FEASIBILITY STUDY on the Use of a DIGITAL PLATFORM for Physical and Psychosocial RECONDITION After Major Neoplastic Surgery
Brief Title: Feasibility Study CORPPS
Acronym: FAISA-CORPPS
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: Santelys Association (Other); ENGIE (Unknown); Fondation Boulanger (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2021_0215; 2021-A02644-37 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2022-05-24; First posted 2022-06-06 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Esophageal Neoplasm; Laryngeal Neoplasms
Keywords: Cancer; Physical and psychosocial rehabilitation; Digital platform; Esophagectomy; Laryngectomy
MeSH Terms: conditions — Esophageal Neoplasms; Laryngeal Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Digital platform — The digital platform consists of 84 exercise sessions of progressive intensity. Each day, the tool offers 8 exercise sessions of about 5 to 10 minutes each, spaced out over an hour. One session can represent several exercises. The patient is asked to perform them daily.

SUMMARY:
The incidence of cancer in France has increased by +135% to reach nearly 400,000 new cases in 2018. The ten-year cancer control strategy 2021-2030 and the health innovation plan have defined strategic axes. Almost all of these axes are addressed in our project. Firstly, the main objective of our study is to improve the quality of life of patients. Secondly, pharyngolaryngeal and oesophageal cancers are among the cancers with a poor prognosis in adults. Thirdly, the project provides access to personalised supportive care for all patients at all times. Finally, the secondary objectives of this study are the prevention of post-operative complications (infectious, thrombo-embolic, pain...).

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized for initial surgical management of esophageal or laryngeal cancer
* Admitted to a conventional ward after partial oesophagectomy or total laryngectomy in a neoplastic setting
* Patient giving consent to participate in the study
* Affiliated to the compulsory health insurance scheme, regardless of the scheme

Exclusion Criteria:

* Patient who did not follow the previously described course of care prior to admission to the ward
* Esophagectomy with total circular pharyngo-laryngectomy
* Total esogastrectomy
* Illiterate, visually impaired patient
* Minor, or adult under guardianship or curatorship, under judicial protection, person deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients hospitalized for surgical management of esophageal or laryngeal cancer in Lille University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2024-04-19 (Actual); Study Completion 2024-04-19 (Actual)

PRIMARY OUTCOMES:
Acceptability rate | At 1 year
  Realization of the ratio between the number of inclusion proposals and the number of accepted inclusions.

SECONDARY OUTCOMES:
Adherence to exercise intervention program: Number of login | Discharge from hospital if it occurs before 30 days or at Day 30
Adherence to exercise intervention program: Number of exercises completed | Discharge from hospital if it occurs before 30 days or at Day 30
Adherence to exercise intervention program: type of exercises completed | Discharge from hospital if it occurs before 30 days or at Day 30
Adherence to exercise intervention program: retention rate | Discharge from hospital if it occurs before 30 days or at Day 30
Satisfaction by the System Usability Scale | Discharge from hospital if it occurs before 30 days or at Day 30
Classification de Clavien-Dindo | At day 30
  Evaluation of the incidence of postoperative complications based on the Clavien-Dindo classification grade II
Visual Analogue Scale | Before and after each activity
  Measure the pain in the scale from 0 to 10
Instant Well-Being Evaluation (IWBE) | Baseline, Discharge from hospital if it occurs before 30 days and at Day 30
  It consists of a graduated scale: the patient must position a cursor, the position on the left corresponding to "I feel very well" and the position on the right to "I do not feel well". The patient is guided by a pictogram (happy, neutral or sad face)
Warwick-Edinburgh Mental Wellbeing Scales | Baseline, Discharge from hospital if it occurs before 30 days and at Day 30
  The well-being and theu quality of life will be assessed using the Warwick-Edinburgh Mental Wellbeing Scales Each item is scored on a range from 1 to 5. The total score will be between 14 and 70, with lower scores indicating poor wellbeing, and higher scores indicating greater wellbeing. Very low wellbeing is defined as a score of ≤ 45. A substantial decrease in wellbeing is a decrease by 5 or more points.
EuroQuol 5 Dimensions (EQ-5D-5L) | Baseline, Discharge from hospital if it occurs before 30 days and at Day 30
  The quality of life will be assessed using the EuroQuol 5 Dimensions The EQ-5D-5L questionnaire will be used to estimate the impact on subjects' health-related quality of life and provides a description of subjects' problems by dimensions (descriptive system), a score for overall self-rated health (visual analogue scale [VAS]) as well as an index score (EQ-5D-5L index). EQ-5D index score range: 0 to 1 and EQ-5D-VAS: range 0 to 100. A higher score indicates better self reported health status.
European Organisation for Research and Treatment of Cancer - Quality of Life Questionnaires (EORTC-QLQ-C30) | Baseline, Discharge from hospital if it occurs before 30 days and at Day 30
  The quality of life will be assessed using the EORTC-QLQ-C30 The Quality of life questionnaire (QLQ-C30) contains 29 items dealing with fatigue, pain, nausea and vomiting, general condition and social, emotional and cognitive functions. It is currently used in many clinical trials in oncology

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume Piessen, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Centre Hospitalier Universtaire, Lille, France